CLINICAL TRIAL: NCT04605744
Title: Implementation of a Peri-procedural Smoking Cessation Program in Patients With Chronic Pain Undergoing Interventional Pain Management Procedures
Brief Title: Peri-procedural Smoking Cessation Program in Patients With Chronic Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the investigators were unable to recruit a sufficient number of participants
Sponsor: The Cooper Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-171
Record Dates: First submitted 2020-10-22; First posted 2020-10-28 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-11

CONDITIONS: Chronic Pain; Smoking
MeSH Terms: conditions — Chronic Pain; Smoking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Smoking cessation counseling — Patients will be given a briefing on the benefits of smoking cessation in the peri-procedural period around their interventional pain procedure. They will also be provided an informational sheet from the American Society of Anesthesiologists promoting cessation. The sheet will contain the 1-800-QUITNOW national hotline phone number.
  Additional an enrollment folder will provided that contains referral information to Cooper's Tobacco Cessation program. This service, free of charge to Cooper Health patients consists of 5 tobacco cessation counselors who use personalized cessation plans, individual and group counseling cessations, Chantix, and education to promote smoking cessation.

SUMMARY:
This single arm study will assess whether smoking cessation counseling offered to chronic pain patients is effective in reducing pain and cigarette use.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Pain of 3 months or greater
* Scheduled for interventional pain procedure

Exclusion Criteria:

* Cancer related pain
* Current participation in smoking abstinence program
* History of schizophrenia or other pyschotic disorder
* History of dementing illness
* Pregnant patients
* Diagnosis of depression or anxiety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Pain | 6 months
  Visual analogue pain score

CONTACTS AND LOCATIONS:
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided